CLINICAL TRIAL: NCT01731405
Title: Consumer Understanding and Use of Medication Guides
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Michael S. Wolf, Associate Professor, Northwestern University
Other Study IDs: ABT-5599; Abbott Laboratories (Other Grant/Funding Number: Abbott Laboratories - 640-5310000-60025599-01)
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Revised Medication Guide Formats
Keywords: Medication Guides; FDA; Prototype; Format

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Formats A,B,C; medicines Ritalin, Morphine Sulfate, Aranesp: All patients will see all 3 different formats of the Medication Guide prototypes. They will also see information for the same drugs, in the same order - Ritalin, Morphine Sulfate, and Aranesp. All participants see all the formats, the only thing that changes by participant is which format is in each medication. There will be 6 different randomized orders - A,B,C; A,C,B; B,C,A; B,A,C; C,A,B; C,B,A. So for example, A,B,C participants would see Ritalin in format A, Morphine Sulfate in format B, and Aranesp in format C.
- There is not another group

SUMMARY:
The purpose of this study is to determine the potential efficacy of three revised Medication Guide layouts to increase consumers' comprehension

DETAILED DESCRIPTION:
'Medication Guides' (Med Guides) are industry-developed documents that have been required by the Food and Drug Administration (FDA) to be issued to consumers for prescription medications that have been viewed to possess "serious and significant public health concerns" since 1998.1,2 These materials for consumers are intended to 1) provide specific dosing administration instructions that could prevent serious adverse effects associated with taking the medication, 2) warn individuals about significant health risks that could affect one's decision to take the medication, or 3) underscore the importance of taking the prescribed medication to the patient's health, and the need for proper adherence.

Despite their potential value in communicating safe and appropriate medication use, problems are clearly evident with the current template for Med Guides. Research conducted by this team in 2006 showed that the majority, if not all Med Guides dispensed with prescribed medicines are too complex and written at a reading grade level not suitable for the majority of patients to comprehend. As a result, these materials are usually ignored by consumers.3 Further research by this team investigating consumers' ability to process and correctly understand content contained in existing Med Guides found that, across all literacy levels, current Med Guides are poorly understood and ineffective in conveying safety information. Patients with low literacy comprehended significantly less, proving yet again that industry standards must be applied to improve these documents.

It is clear that the current guidance for Medication Guide development is insufficient, and the FDA is working to change that. Both the FDA and this research team have proposed multiple new Medication Guide formats, most of which are one-page cover sheets that highlight the most important information of the medication. To examine these new prototypes, this research team conducted six focus groups to obtain consumer-based feedback, and then evaluated three of the prototypes in an eye tracking study. Using the collective data from these two consumer-based studies, the investigators have further developed patient-centered and evidence-based Med Guide prototypes that will be more user-friendly, clear, usable, and low literacy appropriate.

In a cross-sectional, controlled trial, the investigators will investigate consumers' ability to process and correctly understand content contained in each of these top three new, redesigned prototypes.

The purpose of this research is to better understand how well people with varying levels of literacy understand information contained in three newly designed Med Guides. Through an in-person interview, the investigators aim to test consumers' ability to comprehend information contained in the guides by asking them retrieval and inference questions over the guides' content. This will allow us to compare the three formats against each other to see which prototype is most efficient in conveying the important information it is intended to convey. The investigators will recruit a total of 600 participants from general internal medicine clinics here in Chicago (Northwestern clinic = 300 participants and University of Illinois Chicago = 300 participants. A UIC RA will be responsible for this recruitment and will submit their own IRB for review).

This trial will field test our enhanced prototypes and allow us to compare them to each other, showing which format is best understood, especially in participants with low literacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Physically in the primary care clinic

Exclusion Criteria:

* Under 18 years old
* Non-English speaking
* An uncorrectable hearing or a visual impairment which would hinder participants' ability to view the materials
* Too ill to participate
* Moderate to severe cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting from 2 primary care clinics.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Functional Understanding and Comprehension | 30 minute interview
  The primary outcome is to measure which of the three different formats of Medication Guides has the best participant comprehension, which we will assess based on total correct points out of total possible points.

SECONDARY OUTCOMES:
Health Literacy (REALM) | 30 minutes
  The REALM (Rapid Estimate of Adult Health Literacy in Medicine) is a word recognition test designed to provide a valid and quick assessment of participant health literacy.
Participant Characteristics | 30 minutes
  Basic demographic characteristics (age, sex, race/ethnicity), socioeconomic information (education, household income), health status information (self-reported overall health), and recent medication use will be collected by self report.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Wolf, PhD MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Primary Care Plus, Chicago, Illinois

REFERENCES:
- [Background] Tsfasman IM, Starovoitov II, Ziakun AM, Skriabin GK. [Study of the initial reaction of enzymatic oxidation of 1,8-dimethylnaphthalene]. Biokhimiia. 1976 May;41(5):864-8. Russian. PMID 15641
- [Result] Wolf MS, King J, Wilson EA, Curtis LM, Bailey SC, Duhig J, Russell A, Bergeron A, Daly A, Parker RM, Davis TC, Shrank WH, Lambert B. Usability of FDA-approved medication guides. J Gen Intern Med. 2012 Dec;27(12):1714-20. doi: 10.1007/s11606-012-2068-7. Epub 2012 May 8. PMID 22566170
- [Result] Wallace LS, Roskos SE, Weiss BD. Readability characteristics of consumer medication information for asthma inhalation devices. J Asthma. 2006 Jun-Jul;43(5):375-8. doi: 10.1080/02770900600709856. PMID 16801142
- [Result] Safonova TIa, Shelkovskii VI. [Nicotinamide coenzyme level in erythrocytes in children with cerebral paralysis]. Pediatriia. 1977 May;(5):71-3. No abstract available. Russian. PMID 17846
- [Result] Bull C, Goncher G, Deutschman CS, Hoffman BM. Source of residual Bohr effect in hemoglobin oxidation. J Biol Chem. 1977 May 25;252(10):3128-30. PMID 16881
- [Derived] Wolf MS, Bailey SC, Serper M, Smith M, Davis TC, Russell AL, Manzoor BS, Belter L, Parker RM, Lambert B. Comparative effectiveness of patient-centered strategies to improve FDA medication guides. Med Care. 2014 Sep;52(9):781-9. doi: 10.1097/MLR.0000000000000182. PMID 25119953
- See also: Federal Register (FDA-2010-N-0184). Experimental Study of Patient Information Prototypes. — http://edocket.access.gpo.gov/2010/2010-31388.htm